CLINICAL TRIAL: NCT03754179
Title: A lead-in Phase I Followed by a Phase II Clinical Trial on the Combination of Dabrafenib, Trametinib and the Autophagy Inhibitor Hydroxychloroquine in BRAF/MEK Inhibitor-pretreated Patients With Advanced BRAF V600 Mutant Melanoma
Brief Title: Dabrafenib/Trametinib/Hydroxychloroquine for Advanced Pretreated BRAF V600 Mutant Melanoma
Acronym: COMBI-R2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-BN-004
Record Dates: First submitted 2018-11-16; First posted 2018-11-27 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Melanoma
Keywords: autophagy; dabrafenib; hydroxychloroquine; trametinib; melanoma; rechallenge
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A phase 2 (Experimental): Patients are eligible if they are diagnosed with BRAF V600 mutant unresectable AJCC (American Joint Committee on Cancer) stage III or IV melanoma and are documented with progression of disease following treatment with a BRAF with or without MEK inhibitor and treatment with an immune checkpoint inhibitor (at least an anti-PD1 [programmed cell death 1] antibody). Patients will be considered for study participation not earlier than 12 weeks after the last dosing of the prior BRAF with or without MEK inhibitor therapy and 4 weeks after the last dosing of immune checkpoint inhibitor therapy.
  Upfront treatment with dabrafenib 150 mg twice daily, trametinib 2 mg once daily and hydroxychloroquine 200 mg twice daily upfront until disease progression, unacceptable treatment related toxicity or patient's refusal to continue study treatment.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Hydroxychloroquine
- Arm B phase 2 (Active Comparator): Patients are eligible if they are diagnosed with BRAF V600 mutant unresectable AJCC (American Joint Committee on Cancer) stage III or IV melanoma and are documented with progression of disease following treatment with a BRAF with or without MEK inhibitor and treatment with an immune checkpoint inhibitor (at least an anti-PD1 [programmed cell death 1] antibody). Patients will be considered for study participation not earlier than 12 weeks after the last dosing of the prior BRAF with or without MEK inhibitor therapy and 4 weeks after the last dosing of immune checkpoint inhibitor therapy.
  Upfront treatment with dabrafenib 150 mg twice daily, trametinib 2 mg once daily until disease progression. At disease progression, add-on of hydroxychloroquine 200 mg twice daily. Treatment until disease progression, unacceptable treatment related toxicity or patient's refusal to continue study treatment
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Hydroxychloroquine
- Phase 1 (Experimental): Patients are eligible if they are diagnosed with BRAF V600 mutant unresectable AJCC (American Joint Committee on Cancer) stage III or IV melanoma and are documented with progression of disease following treatment with a BRAF with or without MEK inhibitor and treatment with an immune checkpoint inhibitor (at least an anti-PD1 [programmed cell death 1] antibody). Patients will be considered for study participation not earlier than 12 weeks after the last dosing of the prior BRAF with or without MEK inhibitor therapy and 4 weeks after the last dosing of immune checkpoint inhibitor therapy.
  Upfront treatment with dabrafenib 150 mg twice daily, trametinib 2 mg once daily and hydroxychloroquine 200 mg twice daily upfront until disease progression, unacceptable treatment related toxicity or patient's refusal to continue study treatment.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Dabrafenib — Upfront treatment with dabrafenib, trametinib and hydroxychloroquine in phase 1 and Arm A phase 2.
  Upfront treatment with dabrafenib and trametinib in Arm B phase 2 with add-on of hydroxychloroquine at progression of disease
  Other Names: Tafinlar; DAB
Drug: Trametinib — Upfront treatment with dabrafenib, trametinib and hydroxychloroquine in phase 1 and Arm A phase 2.
  Upfront treatment with dabrafenib and trametinib in Arm B phase 2 with add-on of hydroxychloroquine at progression of disease
  Other Names: Mekinist; TRA
Drug: Hydroxychloroquine — Upfront treatment with dabrafenib, trametinib and hydroxychloroquine in phase 1 and Arm A phase 2. Add-on at progression of disease in Arm B phase 2
  Other Names: Plaquenil; HCQ

SUMMARY:
This phase 1/2 trial addresses the efficacy and safety of the combination of dabrafenib, trametinib and the oral autophagy inhibitor hydroxychloroquine in patients with unresectable AJCC (American Joint Committee on Cancer) stage III or stage IV BRAF (v-Raf murine sarcoma viral oncogene homolog B) V600 mutant melanoma who are documented with progression of disease following treatment with a BRAF with or without MEK (MAPK/Erk kinase) inhibitor and treatment with an immune checkpoint inhibitor. The investigators hypothesize hydroxychloroquine will be able to overcome or prevent autophagy-driven resistance to dabrafenib and trametinib. The investigators will also investigate the value of plasma BRAF V600 mutant circulating tumor DNA (ctDNA) as a predictive or prognostic marker.

DETAILED DESCRIPTION:
Lead-in phase 1 safety trial followed by asymmetrically randomized open- label, double-arm, two-stage, multicenter, phase 2 clinical trial.

Patients are eligible if they are diagnosed with BRAF V600 mutant unresectable AJCC (American Joint Committee on Cancer) stage III or IV melanoma and are documented with progression of disease following treatment with a BRAF with or without MEK inhibitor and treatment with an immune checkpoint inhibitor (at least an anti-PD1 [programmed cell death 1] antibody). Patients will be considered for study participation not earlier than 12 weeks after the last dosing of the prior BRAF with or without MEK inhibitor therapy and 4 weeks after the last dosing of immune checkpoint inhibitor therapy.

Phase 1

Patients will be screened and if found eligible treated with the combination of standard dosing of dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) with the autophagy inhibitor hydroxychloroquine (200 mg twice daily). Treatment will continue until disease progression, unacceptable treatment related toxicity or patient's refusal to continue study treatment. Throughout their study participation, patients will be continuously monitored for safety and evaluated for tumor response every 8 weeks or sooner if there is clinical suspicion of progressive disease.

Six patients will be included for this phase 1 trial with incidence of adverse events as primary endpoint and ORR (objective response rate), PFS (progression-free survival), OS (overall survival, per RECIST v1.1 [Response Evaluation Criteria for Solid Tumors]) and value of ctDNA (circulating tumor DNA) as secondary endpoints.

Phase 2

Patients will be screened and if found eligible asymmetrically randomized to treatment with the combination of standard dosing of dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) with the autophagy inhibitor hydroxychloroquine (200 mg twice daily) (arm A, investigational arm) or treatment with standard dosing of dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) (arm B, contemporary control arm). Stratification will occur according to baseline lactate dehydrogenase level. Treatment will continue until disease progression, unacceptable treatment related toxicity or patient's refusal to continue study treatment. However, at disease progression in arm B (dabrafenib plus trametinib), hydroxychloroquine (200 mg twice daily) will be added to the standard treatment and treatment will be continued until disease progression, unacceptable treatment related toxicity or patient's refusal to continue study treatment.

Throughout their study participation, patients will be continuously monitored for safety and evaluated for tumor response every 8 weeks or sooner if there is clinical suspicion of progressive disease.

Primary endpoint is ORR (objective response rate) in arm A, secondary endpoints are ORR (objective response rate) in arm B and PFS (progression-free survival), OS (overall survival), incidence of adverse events and value of ctDNA (circulating tumor DNA) in both arms.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Signed written informed consent.
* Histologically confirmed cutaneous melanoma that is either unresectable AJCC (American Joint Committee on Cancer) stage III or stage IV, and previously determined to be BRAF V600 mutation-positive.
* Subjects must have failed at least two prior systemic anti-cancer treatments for AJCC (American Joint Committee on Cancer) unresectable stage III or stage IV melanoma that must have included: a. Treatment with a BRAF inhibitor (including but not limited to dabrafenib, vemurafenib, encorafenib or other experimental BRAF inhibitors) in combination with a MEK inhibitor (including but not limited to trametinib, cobimetinib, binimetinib or other experimental MEK inhibitors) and progression of disease per Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1 must have been documented during this treatment; b. Treatment with anti-CTLA4 (cytotoxic T-lymphocyt antigen 4) antibodies (ipilimumab or other experimental anti-CTLA4 antibodies), anti-PD1 (programmed cell death 1) antibodies (pembrolizumab, nivolumab or other experimental anti-PD1 antibodies), anti-PDL1 (programmed cell death ligand 1) antibodies and progression of disease per RECIST, version 1.1 or per immune related response criteria must have been documented during this treatment.
* The presence of at least one measurable lesion per RECIST, version 1.1.
* Interval between the date of the last administration of prior therapy for melanoma and the date of recruitment: a. ≥ 12 weeks following the date of the last administration of a BRAF with or without MEK inhibitor; b. ≥ 12 weeks following the date of the first administration and ≥4 weeks following the date of the last administration of ipilimumab, or an anti-PD1, or anti-PD-L1 therapy; c. ≥ 4 weeks following the date of the last administration of chemotherapy (≥ 6 weeks in case of a nitrosurea or mitomycin C containing regimen); d. ≥ 4 weeks following major surgery or extensive radiotherapy.
* All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values as listed on Table 1) must be ≤ grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.0; National Cancer Institute [NCI] 2009) at the time of recruitment.
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to recruitment and agree to use effective contraception throughout the treatment period, and for 16 weeks after the last dose of study treatment.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from 14 days prior to administration of the first dose of study treatment, throughout the treatment period, and for 16 weeks after the last dose of study treatment.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Adequate baseline organ function as defined as follows: Absolute neutrophil count: ≥ 1.2 x 103/mm3 - Hemoglobin: ≥ 9.0 g/dL - Platelet count: ≥ 75 x 103/mm3 - prothrombin time/international normalized ratio and activated partial thromboplastin time: ≤ 1.5 x ULN - Albumin: ≥ 2.5 g/dL - Total bilirubin: ≤ 1.5 x ULN - aspartate aminotransferase and alanine aminotransferase - ≤ 2.5 x ULN - Calculated creatinine clearance - ≥ 50 mL/min (by use of the Cockroft-Gault formula) - Left ventricular ejection fraction ≥ lower limit of normal by transthoracic echocardiogram

Exclusion Criteria:

* No Belgian medical insurance
* Subjects with uveal or mucosal melanoma.
* Prior treatment with hydroxychloroquine, chloroquine or other quinine derivatives.
* Grade 4 or repetitive grade 3 adverse event(s) related to prior treatment with a BRAF and/or a MEK inhibitor.
* Any contra-indication for evaluation by whole body PET/CT (positron emission tomography/computed tomography) and MRI (magnetic resonance imaging) of the brain.
* Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to recruitment.
* Current use of a prohibited medication (macrolides, azoles).
* History of another malignancy with exception of subjects who have been disease-free for 3 years (i.e. subjects with second malignancies that are indolent or definitively treated at least 3 years ago) or subjects with a history of completely resected non-melanoma skin cancer.
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.
* Known Human Immunodeficiency Virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted).
* A history of glucose-6-phosphate dehydrogenase (G6PD) deficiency, psoriasis and/or porphyria.
* No enzyme inducing anticonvulsants for ≥ 4 weeks prior to recruitment.
* A history or evidence of cardiovascular risk including any of the following: a. Current left ventricular ejection fraction < lower limit of normal; b. A QT interval corrected for heart rate using the Bazett's formula (QTcB) ≥480 ms; c. A history or evidence of current clinically significant uncontrolled arrhythmias with exception of subjects with atrial fibrillation controlled for >30 days prior to recruitment are eligible; d. A history (within 6 months prior to recruitment) of acute coronary syndromes (including myocardial infarction or unstable angina), or coronary angioplasty; e. A history or evidence of current ≥ class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines (Appendix 4: New York Heart Association (NYHA) Guidelines); f. Treatment refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by antihypertensive therapy; g. Patients with intra-cardiac defibrillators or permanent pacemakers; h. Known cardiac metastases; i. Abnormal cardiac valve morphology (≥ grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
* Uncorrectable electrolyte abnormalities (e.g. hypokalaemia, hypomagnesaemia, hypocalcaemia), long QT syndrome or taking other medicinal products known to prolong the QT interval.
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including: a. Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); b. Visible retinal pathology as assessed by ophthalmologic examination that is considered a risk factor for RVO or CSR such as: i. Evidence of new optic disc cupping; ii. Evidence of new visual field defects on automated perimetry; iii. Intraocular pressure >21 mmHg as measured by tonography.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
* Females who are nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Ph. 1: incidence of adverse events of DAB, TRA and HCQ | 1 year
  Adverse events graded by the Common Terminology Criteria of Adverse Events version 4 (CTCAE v4)
Ph. 2 Arm A: objective response rate (ORR) of DAB, TRA and HCQ | 2 years
  Objective response rate (ORR; defined as the percentage of subjects with a confirmed complete response [CR] or partial response [PR] at any time per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1 [Eisenhauer 2009]).

SECONDARY OUTCOMES:
Ph. 1: objective response rate (ORR) of DAB, TRA and HCQ | 1 year
  Objective response rate (ORR; defined as the percentage of subjects with a confirmed complete response [CR] or partial response [PR] at any time per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1 [Eisenhauer 2009]).
Ph. 1: progression-free survival (PFS) on DAB, TRA and HCQ | 1 year
  Progression-free survival (PFS; defined as the time from treatment initiation until the earliest date of disease progression or death due to any cause)
Ph. 1: overall survival (OS) on DAB, TRA and HCQ | 1 year
  Overall survival (OS; defined as the time from treatment initiation until the date of death due to any cause).
Ph. 1: value of BRAF V600 mutant circulating tumor DNA (ctDNA) as a predictive and/or prognostic marker during treatment DAB, TRA and HCQ | 1 year
  Copy number of BRAF V600 mutant ctDNA as measured by quantitative Polymerase Chain Reaction (qPCR)
Ph. 2 Arm B: objective response rate 1 (ORR 1) of DAB and TRA prior to the addition of HCQ at progression of disease | 2 years
  Objective response rate 1 (ORR 1; defined as the percentage of subjects with a confirmed complete response [CR] or partial response [PR] prior to the addition of hydroxychloroquine at any time per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1 [Eisenhauer 2009]).
Ph. 2 Arm B: objective response rate 2 (ORR 2) of DAB and TRA following the addition of HCQ at progression of disease | 2 years
  Objective response rate 2 (ORR 2; defined as the percentage of subjects with a confirmed complete response [CR] or partial response [PR] following the addition of hydroxychloroquine at any time per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1 [Eisenhauer 2009]).
Ph. 2 Arm A: progression-free survival (PFS) on DAB, TRA and HCQ | 2 years
  Progression-free survival (PFS; defined as the time from randomization until the earliest date of disease progression or death due to any cause)
Ph. 2 Arm A: overall survival (OS) on DAB, TRA and HCQ | 2 years
  Overall survival (OS; defined as the time from randomization until the date of death due to any cause).
Ph. 2 Arm B: progression-free survival 1 (PFS 1) on DAB and TRA prior to the addition of HCQ | 2 years
  Progression-free survival 1 (PFS 1; defined as the time from randomization until the earliest date of disease progression or death due to any cause whilst treated with dabrafenib and trametinib)
Ph. 2 Arm B: progression-free survival 2 (PFS 2) on DAB and TRA following the addition of HCQ | 2 years
  Progression-free survival 2 (PFS 2; defined as the time from addition of hydroxychloroquine to dabrafenib and trametinib until the earliest date of disease progression or death due to any cause)
Ph. 2 Arm B: overall survival 1 (OS 1) on DAB and TRA prior to the addition of HCQ | 2 years
  Overall survival 1 (OS 1; defined as the time from randomization until death due to any cause whilst treated with dabrafenib and trametinib)
Ph. 2 Arm B: overall survival 2 (OS 2) on DAB and TRA following the addition of HCQ | 2 years
  Overall survival 2 (OS 2; defined as the time from addition of hydroxychloroquine to dabrafenib and trametinib until death due to any cause)
Ph. 2 Arm B: overall survival 3 (OS 3) on DAB and TRA following the addition of HCQ | 2 years
  Overall survival 3 (OS 3; defined as the time from randomization until death).
Ph. 2 Arm A and B: incidence of adverse events of DAB, TRA and HCQ | 2 years
  Adverse events graded by the Common Terminology Criteria of Adverse Events version 4 (CTCAE v4)
Ph. 2 Arm A and B: value of BRAF V600 mutant circulating tumor DNA (ctDNA) as a predictive and/or prognostic marker during treatment with DAB, TRA and HCQ | 2 years
  Copy number of BRAF V600 mutant ctDNA as measured by quantitative Polymerase Chain Reaction (qPCR) in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided